CLINICAL TRIAL: NCT04156178
Title: Phase I, Interventional, Single Arm, Open Label, Treatment Study to Evaluate the Safety and Tolerability of CD20-CD19 cCAR in Patients With Relapsed and/or Refractory B Cell Malignancies
Brief Title: CD20-CD19 Compound CAR (cCAR) T Cells for Patients With Relapsed /Refractory B Cell Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: Peking University Shenzhen Hospital (Other); Chengdu Military General Hospital (Other); iCAR Bio Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICG133-001
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-01

CONDITIONS: B Cell Lymphoma; B Cell Leukemia
Keywords: CD20; CD19; cCAR; Leukemia; Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell; Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD20-CD19 cCAR T cells (Experimental): CD20-CD19 cCAR T cells transduced with a lentiviral vector to express two distinct units of anti-CD20 and CD19 CARs
  Interventions: Biological: CD20-CD19 cCAR T cells

INTERVENTIONS:
Biological: CD20-CD19 cCAR T cells — CD20-CD19 cCAR T cells administered to patients, will be either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of CD20-CD19 cCAR in patients with relapsed and/or refractory B cell malignancies.

DETAILED DESCRIPTION:
Clinical trials with CD19-directed CARs have achieved unprecedented remission rates as high as 90%. However, recent follow-up studies have shown a substantial portion of treated patients relapsed due to antigen escape. CD20-CD19 cCAR is a compound Chimeric Antigen Receptor (cCAR) immunotherapy with two distinct functional CAR molecules expressed on a T-cell, directed against the surface proteins CD20 and CD19. CD20-CD19 cCAR intends to target the mechanisms of single-CAR relapse, specifically antigen escape.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis based on the World Health Organization (WHO) 2008
2. Histologically demonstrate CD19 or CD20 expressing B cell lymphoma or B ALL
3. Patients have exhausted standard therapeutic options
4. Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks
5. Female must be not pregnant during the study

Exclusion Criteria:

1. Patients declining to consent for treatment
2. Prior solid organ transplantation
3. Potentially curative therapy including chemotherapy or hematopoietic cell transplant
4. Prior treatment with CD20xCD3 or CD19x3 bispecific agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 28 days
Type of dose-limiting toxicity (DLT) | 28 days
Number of participants with adverse event by severity as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 2 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  Assessment of morphologic complete remission (CR), complete remission with incomplete recovery of counts (CR1), no residual disease as analyzed by flow cytometry analysis, and molecular remission by molecular studies
Progression-free survival (PFS) | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhang, MD, PhD, Principal Investigator — Peking University Shenzhen Hospital; Fang Liu, MD, PhD, Principal Investigator — Chengdu Military General Hospital
Locations (2):
- China (2):
  - Chengdu Military General Hospital, Chengdu
  - Peking University Shenzhen Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No